CLINICAL TRIAL: NCT04715919
Title: Long Term Outcomes in Patients With Coronavirus Disease-19 (COVID-19) on Pulmonary Functions, Exercise Capacity, Lung Structure and Quality of Life
Brief Title: Long Term Outcomes of Coronavirus Disease-19 (COVID-19)
Status: Completed | Type: Observational
Sponsor: Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital (Other)
Collaborators: Turkish Respiratory Society (Unknown)
Responsible Party: Principal Investigator, Cenk Kirakli, M.D., Professor Doctor, Izmir Dr Suat Seren Chest Diseases and Surgery Education and Research Hospital
Other Study IDs: 195/ADF14
Record Dates: First submitted 2020-12-28; First posted 2021-01-20 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Covid19
Keywords: Covid19; Long term outcomes; Chest computed comography; Pulmonary functional tests; Exercise capacity; Quality of life
MeSH Terms: conditions — COVID-19 | interventions — Respiratory Function Tests; Quality of Life

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients in ICU: ICU patients with COVID-19
  Interventions: Diagnostic Test: Chest Computed Tomography; Diagnostic Test: Pulmonary Function Tests; Other: Six Minutes Walk Test; Other: Quality of Life
- Patients in Hospital Ward: Patients with COVID-19 in hospital wards
  Interventions: Diagnostic Test: Chest Computed Tomography; Diagnostic Test: Pulmonary Function Tests; Other: Six Minutes Walk Test; Other: Quality of Life

INTERVENTIONS:
Diagnostic Test: Chest Computed Tomography — Evaluation of Lung Structure
Diagnostic Test: Pulmonary Function Tests — Respiratory Capacity
Other: Six Minutes Walk Test — Exercise Capacity
Other: Quality of Life — Physical disability assessment tool
  Other Names: SF-36

SUMMARY:
The investigators hypothese that lung involvement due to COVID-19 may cause structural changes in the lung in the long term. In this study the effects of structural changes in the lung on pulmonary function tests, exercise capacity and quality of life will be examined.

DETAILED DESCRIPTION:
Coronavirus disease-19 (COVID-19) has a clinical spectrum ranging from asymptomatic cases to severe cases requiring intensive care hospitalization due to respiratory failure. The disease mostly infects the lower respiratory tract. Typical computed tomography findings of lung involvement are bilateral, peripherally located ground glass density and consolidations. There is a close relationship between tomography findings and clinical severity. It is not known whether there will be complete recovery in the lungs.

Investigators will evaluate pulmonary structures with chest computed tomography, respiratory capacity with pulmonary function tests (PFTs), exercise capacity with six minutes walk test and quality of life with short form-36 (SF-36) im patients who survivors of COVID-19 at least 6 months after hospital discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were ≥18 years
* COVID-19 confirmed by Real-Time PCR
* At least 6 months after discharge

Exclusion Criteria:

* Patients who were < 18 years
* Pregnancy
* Become bedridden after discharge

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Survivors of COVID-19 aged over 18 years old who had been admitted in University of Health Sciences, Dr. Suat Seren Chest Disease and Surgery Training and Research Hospital for COVID-19 patients in İzmir, Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
Structural Change in Lung | up to 6 months after discharge
  Chest Computed Tomography

SECONDARY OUTCOMES:
Carbon monoxide diffusion capacity (DLCO) | up to 6 months after discharge
  Carbon monoxide diffusion capacity of the lung
Exercise Capacity | up to 6 months after discharge
  Six Minutes Walking Test
Short Form Health Survey Score (SF-16) | up to 6 months after discharge
  A 36-item patient-reported questionnaire that covers eight health domains: physical functioning (10 items), bodily pain (2 items), role limitations due to physical health problems (4 items), role limitations due to personal or emotional problems (4 items), emotional well-being (5 items), social functioning (2 items), energy/fatigue (4 items), and general health perceptions (5 items). Scores for each domain range from 0 to 100, with a higher score defining a more favorable health state

CONTACTS AND LOCATIONS:
Locations (1):
- 1University of Health Sciences Turkey, Dr Suat Seren Chest Diseases and Chest Surgery Training and Research Hospital, Intensive Care Unit, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No